CLINICAL TRIAL: NCT04689568
Title: Improving Depression Via E-Health Access (IDEA) Study: Evaluating Uptake and Efficacy of Self-Help e-Mental Health Interventions in Primary Care
Brief Title: Improving Depression Via E-Health Access (IDEA) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jennifer Severe, Assistant Professor of Psychiatry, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00174081
Record Dates: First submitted 2020-12-27; First posted 2020-12-30 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: This is a single-center, non-randomized, preferred assignment study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moodkit (Active Comparator): MoodKit is a cognitive behavioral therapy (CBT)-based app designed to provide tools for managing depressed mood, anxiety and stress.
  Interventions: Behavioral: Moodkit
- Moodgym (Active Comparator): Moodgym is an online cognitive behavioral therapy (CBT)-based program designed to prevent or reduce symptoms of depression and anxiety by helping users identify and overcome problem emotions and to develop good coping skills.
  Interventions: Behavioral: Moodgym
- University of Michigan Depression Center Toolkit (Active Comparator): The Toolkit provides information, tools, support, and resources to guide individuals through their mental health journey. The Toolkit offers help to people who are experiencing problems with a mood disorder as well as with stress and anxiety.
  Interventions: Behavioral: University of Michigan Depression Center Toolkit

INTERVENTIONS:
Behavioral: Moodkit — MoodKit is divided into four main sections: Activities, Thoughts, Mood and Journal. In the Thoughts section, the user is asked to briefly describe stressful situations and their reactions to the event and is later educated on a number of "thought distortions". In the Mood section, the user is asked to give an overall rating of mood, which can be done several times per day. In the Journal section, the user can write freestanding journal entries. Additional areas of advice and goal setting are contained in a section called Thrive Tips.
  Arms: Moodkit
Behavioral: Moodgym — The program consists of five modules each taking 20- to 40-minutes to complete, which are completed in a prescribed order.
  Arms: Moodgym
Behavioral: University of Michigan Depression Center Toolkit — The Toolkit provides information, tools, support, and resources to guide individuals through their mental health journey.
  Arms: University of Michigan Depression Center Toolkit

SUMMARY:
The researchers are doing this study to learn more about which online self-help resources, including a smartphone app, an online program, or an informational website, primary care patients with depression are likely to choose and whether the chosen tool will improve their depressive symptoms and wellbeing. The researchers would also like to know how likely someone is to use the resources and their satisfaction with the resources.

DETAILED DESCRIPTION:
Participants will be using a self-help resource for the 6-week study period. A Care Manager will contact participants by phone, once a week, for about 5-10 minutes at a pre-arranged time. Participation will be needed for 10 weeks in total (6 weeks of active participation and a survey 1-month after the study intervention ends).

Subscription-based self-help resources being tested during the study will not be freely available after the study period. However, the researchers will share information on how to access these resources for a fee after the study period to all participants.

In addition to the time above, the researchers will collect information from participant's medical records for another 10 months after participation. The entire study is expected to last about 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are English-speaking
* Individuals with a Patient Health Questionnaire 9 (PHQ9) score greater than or equal to 11 or diagnosis of moderate to severe depression determined by the Care Manager during her initial psychiatric evaluation and by the study PI during panel review will supersede a low PHQ9 score.
* Individuals with have daily internet access and a smartphone;
* Individuals who agree to periodic contact with the care manager and study team.

Exclusion Criteria:

* Individuals who have cognitive impairment that would preclude use of self-help resources
* Individuals with already using an electronic mental health resource;
* Individuals with unstable medical illness, e.g. active cancer;
* Individuals with severe psychiatric symptoms (marked suicidality, psychotic symptoms, severe substance abuse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Patient preference, use and satisfaction of the intervention as assessed by timed structured survey | Up to 14 months
Patient frequency and duration of intervention use and satisfaction as assessed by weekly structured survey | Up to 14 months
  Structured survey conducted weekly.
Patient preference and satisfaction with the intervention as assessed by qualitative interviews | Up to approximately 14 months
  Interviews are semi-structured and audio recorded
Care manager experiences of the intervention as assessed by qualitative interviews | Up to approximately 18 months
  Interviews are semi-structured and audio recorded
Clinician/Administrator views related to interventions as assessed by qualitative interviews | Up to approximately 18 months
  Interviews are semi-structured and audio recorded
Patient frequency of intervention use as assessed by self-report use of tools | Up to 14 months
  As recorded in participants' printed copy of their mood-logs from the app or program.
Change in severity of symptoms of depression as assessed with the Patient Health Questionnaire 9 (PHQ-9) score | At baseline (before choosing an intervention) and at week 6 (when they complete the intervention)
  The PHQ-9 is an instrument for screening, diagnosing, monitoring and measuring the severity of depression: The PHQ-9 has a range of scores from 0-27. Depression Severity: 0- none, 1-4 minimal, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Change in level of functioning as assessed with the Sheehan Disability Scale (SDS) | At baseline (before choosing an intervention) and at week 6 (when they complete the intervention)
  The Sheehan Disability Scale (SDS) is a 5-item clinician-rated questionnaire used to evaluate impairments in the domains of work, social life/leisure, and family life/home responsibility. All items are rated on a continuum (0 = no impairment to 10 = most severe) with the total SDS score ranging from 0 (no impairment) to 30 (most severe)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Severe, MD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No